CLINICAL TRIAL: NCT04389723
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Investigate the Safety and Efficacy of Qualia Mind on Cognition in a Healthy Population
Brief Title: Safety and Efficacy Study of Qualia Mind on Cognition in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurohacker Collective (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 20QCHN
Record Dates: First submitted 2020-04-30; First posted 2020-05-15 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Healthy; Cognitive Function
Keywords: Cognition; Nootropic; Dietary Supplement; Healthy; Cambridge Brain Science Test

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo→ Qualia Mind (Other): Subjects are first administered the placebo then crossover to the investigational product
  Interventions: Dietary Supplement: Qualia Mind; Dietary Supplement: Placebo
- Qualia Mind→ Placebo (Other): Subjects are first administered the investigational product then crossover to the placebo
  Interventions: Dietary Supplement: Qualia Mind; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Qualia Mind — Multi-ingredient Dietary supplement
Dietary Supplement: Placebo — Multi-ingredient Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, crossover study designed to investigate the safety and efficacy of Qualia Mind on cognition in a healthy adult population between ages of 18 and 75 years. Qualia Mind is a nootropic supplement containing a complex mixture of vitamins, minerals, amino acids, choline donors, and herbal ingredients. These components have been demonstrated to exert their cognitive effects through distinct mechanisms of action involving cholinergic, glutamatergic, and dopaminergic receptor signalling; neuroplasticity; and modulation of cell membrane structure and metabolism.

DETAILED DESCRIPTION:
Qualia Mind is a nootropic supplement containing a complex mixture of vitamins, minerals, amino acids, choline donors, and herbal ingredients. These components have been demonstrated to exert their cognitive effects through distinct mechanisms of action involving cholinergic, glutamatergic, and dopaminergic receptor signalling; neuroplasticity; and modulation of cell membrane structure and metabolism. Vitamin B6 and B12 supplementation have been shown to improve cognitive scores related to memory in healthy participants aged 20 to 92 years. Twenty-eight days of B vitamin complex and vitamin C supplementation increased subjective ratings of concentration, mental stamina, and alertness. Although each B vitamin may exert differential effects on cognition, a higher intake of B vitamins throughout adulthood is associated with greater cognitive function later in life. An acute dose of CDP-choline improved processing speed, memory, verbal learning, and executive functioning in healthy participants who were poor performers on tests at baseline. Cognitive improvement among all participants may have been observed with repeated administration. It is also expected that with the additional administration of uridine monophosphate (UMP) and docosahexaenoic acid (DHA), a long-chain polyunsaturated fatty acid, would have a greater effect on cognitive performance based on preclinical studies describing a synergistic effect between the ingredients. Phosphatidylserine (PS) daily supplementation has strong clinical support for use in healthy humans for enhancing cognition and maintaining cognitive baseline performance. Moreover, the cognitive effects of Ginkgo biloba were found to be superior when complexed with PS. A specific extract of the herbal adaptogen, Bacopa monnieri, prepared from stems, leaves, and roots of the plant has been shown in healthy populations to enhance cognition by improving memory recall, selective attention, and processing speed. Rhodiola rosea, another herbal adaptogen, improved speed, and accuracy, compared to placebo, in a choice reaction time task using an extract derived from roots of the plant following a 4-week supplementation period. Examination of individual and synergistic effects of theobromine and caffeine in preclinical and clinical studies have been generally positive. Several doses of theobromine with caffeine have been shown to improve alertness, working memory, and other cognitive facets. Caffeine in combination with L-theanine has also been demonstrated to improve processing speed and accuracy in an attention-switching task, while improving concentration in a memory task. Other ingredients, such as Celastrus paniculatus, and pyrroloquinoline quinone have preclinical evidence supporting their positive effect on cognition that warrants further investigations in the form of clinical trials.

A previous open-label study in a healthy population consuming Qualia Mind for 5 days assessed cognition using the Cambridge Brain Science Test and found significant improvements in memory, concentration, reasoning, and planning skills compared to baseline. Participants reported a significant 85% improvement in concentration after 5 days of supplementation. These promising preliminary results, however, require placebo-controlled studies to aid their interpretation.

While the interest in enhancing cognitive performance is growing along with the use of brain health supplements, it is important to establish the safety and efficacy of nootropic supplements. Prescription and prohibited stimulant drugs intended to enhance mental performance have been increasing in usage worldwide. In 2017, results from the Global Drug Survey found that 14% of respondents reported using stimulants at least once in the last 12 months, an increase from the 5% reported in the previous year. In the US alone, the use of drugs specifically for cognitive enhancement rose from 20 to 30%. These individuals seeking out cognitive enhancement primarily used prescription drugs, that are designed for individuals with Attention Deficit Hyperactivity Disorder (ADHD), such as the popular methylphenidate (Ritalin) or amphetamine-dextroamphetamine (Adderall).

However, the evidence that these drugs enhance cognition in individuals without ADHD is lacking. Moreover, the misuse of stimulants is associated with adverse effects, such as psychosis, anorexia, cardiovascular events, and sudden death. The alternative nootropic industry of cognitive enhancers is a safe and legal substitute, with supplements designed specifically for healthy individuals. It is likely that stimulant misuse and associated adverse effects will be reduced, with the growing popularity and availability of clinically proven nootropics.

Based on the existing evidence on individual ingredients and preliminary studies on Qualia Mind, the current randomized, double-blind, placebo-controlled, crossover study is designed to investigate the safety and efficacy of Qualia Mind on cognition in a healthy adult population between ages of 18 and 75 years.

ETHICAL ASPECTS OF THE STUDY

This study will be conducted with the highest respect for the individual participants (i.e., participants) according to the protocol, the ethical principles that have their origin in the Declaration of Helsinki, and the ICH Harmonised Tripartite Guideline for GCP.

STATISTICAL EVALUATION

Analysis Plan

The Safety Population will consist of all participants who received any amount of either product and on whom any post-randomization safety information is available.

The Intent-to-Treat (ITT) Population consists of all participants who received either product and on whom any post-randomization efficacy information is available.

The Per Protocol (PP) Population consists of all participants who consumed at least 80% of treatment or placebo doses, do not have any major protocol violations and complete all study visits and procedures connected with measurement of the primary variable.

Statistical Analysis Plan

All hypothesis testing will be carried out at the 5% (2-sided) significance level unless otherwise specified.

All data will be summarised by study group and/or visit. For continuous variables, the minimum and maximum, the arithmetic mean, median and standard deviation will be presented to two decimal places. For categorical variables, counts and percentages will be described. The denominator for each percentage will be the number of subjects within the population study group unless otherwise specified.

The formula for the changes of continuous endpoints from screening/baseline:

Change to Vi = Value at Vi - Value at V screening/baseline For the primary outcomes, analysis of covariance (ANCOVA) will be conducted for the evaluation of the change from baseline to the follow-up visit. The model will include period, group and sequence as fixed effects.

ELIGIBILITY:
Inclusion Criteria:

1. Provided voluntary, written, informed consent to participate in the study
2. Male and female participants between 18 and 75 years of age, inclusive
3. BMI between 18.5 to 32.5 kg/m2, inclusive
4. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices (implanted for at a minimum of 3 months)
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
5. Men must agree to the use of condoms unless partner is using an acceptable form of female contraception as defined in inclusion #4 during the study period and for at least 7 days after completion of the study
6. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
7. A score of ≥ 25 on MMSE-2 (Section 9.7.5)
8. Agrees to avoid high caffeine consumption starting 5-days prior to visit 2 and during the study (equivalent to no more than 2 standard cups of caffeinated coffee or tea per day)
9. Agrees to avoid caffeine consumption 24 hours prior to in-clinic visits
10. Agrees to avoid alcohol consumption 24 hours prior to in-clinic visits
11. Agrees to avoid cannabis use 24 hours prior to in-clinic visits
12. Have a regular sleep-wake cycle with a bedtime between 9:00 pm and 12:00 am and receive between 7 and 9 hours of sleep for at least 3 weeks prior to baseline
13. Agrees to maintain current sleep schedule throughout study
14. Agrees to maintain current level of physical activity and diet throughout the study
15. Healthy as determined by medical history and laboratory results as assessed by QI

Exclusion Criteria:

1. Individuals who are cognitively impaired and/or who are unable to give informed consent
2. Women who are pregnant, breastfeeding or planning to become pregnant during the trial
3. Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients
4. Previous diagnosis of a sleep disorder
5. Currently experiencing vivid nightmares or sleepwalking
6. Current employment that calls for rotating shift work or shift work that will disrupt normal circadian rhythm in the last 3 weeks
7. Unstable metabolic disease or chronic diseases as assessed by the QI
8. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
9. Type I or Type II diabetes
10. A significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case by case basis
11. Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Participants with minor surgery will be considered on a case-by-case basis by the QI
12. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
13. Individuals with an autoimmune disease or are immune-compromised
14. Self-reported diagnosis of HIV-, Hepatitis B- and/or C-positive
15. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom-free for 6 months
16. Self-reported current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
17. Self-reported medical or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation
18. Current or history of any significant diseases of the gastrointestinal tract
19. Blood/bleeding disorders as determined by laboratory results
20. Current use of prescribed medications listed in the protocol
21. Current use of over-the-counter medications, supplements, foods and/or drinks listed in the protocol
22. Chronic use of cannabinoid products (>2 times/week)
23. Use of tobacco products within 60 days of the baseline visit and during the study period
24. Self-reported alcohol or drug abuse within the last 12 months
25. Self-reported high alcohol intake (average of >2 standard drinks per day or >10 standard drinks per week)
26. Clinically significant abnormal laboratory results at screening as assessed by the QI
27. Blood donation 30 days prior to screening, during the study, or a planned donation within 30-days of the last study visit
28. Participation in other clinical research trials 30 days prior to screening
29. Any other condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
The difference in the change from baseline in Overall Mental Performance after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Combined Verbal Ability scores after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Combined Reasoning Scores after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.

SECONDARY OUTCOMES:
The difference in the change from baseline in combined Short-term Memory Scores after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Verbal Reasoning after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Deductive Reasoning after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Alternating Attention after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Selective Attention after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Planning after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Verbal Short-Term Memory after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Spatial Short- Term Memory after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Episodic Memory after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Spatial Memory after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Working Memory after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Visuospatial Working Memory after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.
The difference in the change from baseline in Visuospatial processing after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Assessed using Cambridge Brain Science Test comprising a total of 12 assessments, each of which is a neurocognitive task that measures a core element of cognition. Four cognitive domains Overall Mental Performance, Verbal Ability, Reasoning and Short-term Memory scores will be calculated from using scores from the 12 assessments. Based on previous studies (1), these scores may range from -3.70 to 4.01 or beyond. Scores greater than 0 are above average and those less than 0 are below average. Scores for individual assessments may range from -39 through 240 or beyond.

OTHER OUTCOMES:
Incidence of pre-emergent adverse eventsafter 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Incidence of post-emergent adverse events after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in systolic blood pressure after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in diastolic blood pressure after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in heart rate after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood alanine aminotransferase (ALT) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood creatinine after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood aspartate transaminase (AST) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood total bilirubin after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood sodium (Na) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood potassium (K) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood chloride (Cl) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood glucose after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in blood estimated glomerular filtration rate (eGFR) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in white blood cell (WBC) count after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in neutrophils after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in lymphocytes after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in monocytes after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in eosinophils after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in basophils after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in red blood cell (RBC) count after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in hemoglobin after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
Change in hematocrit after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Parameters to be assessed are: white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV))
Change in platelet count after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Parameters to be assessed are: white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV))
Change in mean corpuscular volume (MCV) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Parameters to be assessed are: white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV))
Change in mean corpuscular hemoglobin (MCH) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Parameters to be assessed are: white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV))
Change in mean corpuscular hemoglobin concentration (MCHC) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Parameters to be assessed are: white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV))
Change in red cell distribution width (RDW) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Parameters to be assessed are: white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV))
Change in mean platelet volume (MPV) after 5 days of supplementation with Qualia Mind compared to placebo | 5 days
  Parameters to be assessed are: white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV))

CONTACTS AND LOCATIONS:
Overall Officials: Rupal Trivedi, MD, Principal Investigator — Great Lakes Clinical Trials LLC
Locations (1):
- Great Lakes Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manders M, de Groot LC, van Staveren WA, Wouters-Wesseling W, Mulders AJ, Schols JM, Hoefnagels WH. Effectiveness of nutritional supplements on cognitive functioning in elderly persons: a systematic review. J Gerontol A Biol Sci Med Sci. 2004 Oct;59(10):1041-9. doi: 10.1093/gerona/59.10.m1041. PMID 15528776
- [Background] Kennedy DO, Veasey RC, Watson AW, Dodd FL, Jones EK, Tiplady B, Haskell CF. Vitamins and psychological functioning: a mobile phone assessment of the effects of a B vitamin complex, vitamin C and minerals on cognitive performance and subjective mood and energy. Hum Psychopharmacol. 2011 Jun-Jul;26(4-5):338-47. doi: 10.1002/hup.1216. Epub 2011 Jul 12. PMID 21751253
- [Background] Qin B, Xun P, Jacobs DR Jr, Zhu N, Daviglus ML, Reis JP, Steffen LM, Van Horn L, Sidney S, He K. Intake of niacin, folate, vitamin B-6, and vitamin B-12 through young adulthood and cognitive function in midlife: the Coronary Artery Risk Development in Young Adults (CARDIA) study. Am J Clin Nutr. 2017 Oct;106(4):1032-1040. doi: 10.3945/ajcn.117.157834. Epub 2017 Aug 2. PMID 28768650
- [Background] Knott V, de la Salle S, Choueiry J, Impey D, Smith D, Smith M, Beaudry E, Saghir S, Ilivitsky V, Labelle A. Neurocognitive effects of acute choline supplementation in low, medium and high performer healthy volunteers. Pharmacol Biochem Behav. 2015 Apr;131:119-29. doi: 10.1016/j.pbb.2015.02.004. Epub 2015 Feb 12. PMID 25681529
- [Background] Holguin S, Martinez J, Chow C, Wurtman R. Dietary uridine enhances the improvement in learning and memory produced by administering DHA to gerbils. FASEB J. 2008 Nov;22(11):3938-46. doi: 10.1096/fj.08-112425. Epub 2008 Jul 7. PMID 18606862
- [Background] Glade MJ, Smith K. Phosphatidylserine and the human brain. Nutrition. 2015 Jun;31(6):781-6. doi: 10.1016/j.nut.2014.10.014. Epub 2014 Nov 4. PMID 25933483
- [Background] Kennedy DO, Haskell CF, Mauri PL, Scholey AB. Acute cognitive effects of standardised Ginkgo biloba extract complexed with phosphatidylserine. Hum Psychopharmacol. 2007 Jun;22(4):199-210. doi: 10.1002/hup.837. PMID 17457961
- [Background] Benson S, Downey LA, Stough C, Wetherell M, Zangara A, Scholey A. An acute, double-blind, placebo-controlled cross-over study of 320 mg and 640 mg doses of Bacopa monnieri (CDRI 08) on multitasking stress reactivity and mood. Phytother Res. 2014 Apr;28(4):551-9. doi: 10.1002/ptr.5029. Epub 2013 Jun 21. PMID 23788517
- [Background] Pase MP, Kean J, Sarris J, Neale C, Scholey AB, Stough C. The cognitive-enhancing effects of Bacopa monnieri: a systematic review of randomized, controlled human clinical trials. J Altern Complement Med. 2012 Jul;18(7):647-52. doi: 10.1089/acm.2011.0367. Epub 2012 Jul 2. PMID 22747190
- [Background] Jowko E, Sadowski J, Dlugolecka B, Gierczuk D, Opaszowski B, Cieslinski I. Effects of Rhodiola rosea supplementation on mental performance, physical capacity, and oxidative stress biomarkers in healthy men. J Sport Health Sci. 2018 Oct;7(4):473-480. doi: 10.1016/j.jshs.2016.05.005. Epub 2016 May 20. PMID 30450257
- [Background] Cova I, Leta V, Mariani C, Pantoni L, Pomati S. Exploring cocoa properties: is theobromine a cognitive modulator? Psychopharmacology (Berl). 2019 Feb;236(2):561-572. doi: 10.1007/s00213-019-5172-0. Epub 2019 Jan 31. PMID 30706099
- [Background] Owen GN, Parnell H, De Bruin EA, Rycroft JA. The combined effects of L-theanine and caffeine on cognitive performance and mood. Nutr Neurosci. 2008 Aug;11(4):193-8. doi: 10.1179/147683008X301513. PMID 18681988
- [Background] Ohwada K, Takeda H, Yamazaki M, Isogai H, Nakano M, Shimomura M, Fukui K, Urano S. Pyrroloquinoline Quinone (PQQ) Prevents Cognitive Deficit Caused by Oxidative Stress in Rats. J Clin Biochem Nutr. 2008 Jan;42(1):29-34. doi: 10.3164/jcbn.2008005. PMID 18231627
- [Background] Bhanumathy M, Harish MS, Shivaprasad HN, Sushma G. Nootropic activity of Celastrus paniculatus seed. Pharm Biol. 2010 Mar;48(3):324-7. doi: 10.3109/13880200903127391. PMID 20645820
- [Background] Pan X, Gong N, Zhao J, Yu Z, Gu F, Chen J, Sun X, Zhao L, Yu M, Xu Z, Dong W, Qin Y, Fei G, Zhong C, Xu TL. Powerful beneficial effects of benfotiamine on cognitive impairment and beta-amyloid deposition in amyloid precursor protein/presenilin-1 transgenic mice. Brain. 2010 May;133(Pt 5):1342-51. doi: 10.1093/brain/awq069. Epub 2010 Apr 12. PMID 20385653
- [Background] Maier LJ, Ferris JA, Winstock AR. Pharmacological cognitive enhancement among non-ADHD individuals-A cross-sectional study in 15 countries. Int J Drug Policy. 2018 Aug;58:104-112. doi: 10.1016/j.drugpo.2018.05.009. Epub 2018 Jun 11. PMID 29902691
- [Background] Lakhan SE, Kirchgessner A. Prescription stimulants in individuals with and without attention deficit hyperactivity disorder: misuse, cognitive impact, and adverse effects. Brain Behav. 2012 Sep;2(5):661-77. doi: 10.1002/brb3.78. Epub 2012 Jul 23. PMID 23139911
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Hampshire A, Highfield RR, Parkin BL, Owen AM. Fractionating human intelligence. Neuron. 2012 Dec 20;76(6):1225-37. doi: 10.1016/j.neuron.2012.06.022. PMID 23259956
- [Background] Wild CJ, Nichols ES, Battista ME, Stojanoski B, Owen AM. Dissociable effects of self-reported daily sleep duration on high-level cognitive abilities. Sleep. 2018 Dec 1;41(12):zsy182. doi: 10.1093/sleep/zsy182. PMID 30212878
- See also: Pilot study: Qualia Mind: Neurohacker Collective — https://neurohacker.com/qualia-mind-pilot-study?inf_contact_key=bd86be8af5addb3500976a70cff578a04dfbc39d7283b2cb89d5189540b69330
- See also: Use of 'smart drugs' on the rise — https://www.nature.com/articles/d41586-018-05599-8